CLINICAL TRIAL: NCT06755983
Title: The Effect of Endorphin Massage Applied Before Mastectomy Surgery on Surgical Fear, Anxiety and Pain Levels
Brief Title: Effect of Endorphin Massage on Surgical Fear, Anxiety and Pain Before Mastectomy
Acronym: Mastectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, MERVE KAYA, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MERVE KAYA
Record Dates: First submitted 2024-12-18; First posted 2025-01-01 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Pain; Anxiety; Fear
Keywords: mastectomy; pain; anxiety; fear; endorphin massage
MeSH Terms: conditions — Pain, Postoperative; Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endhorphin massage grup (Experimental): The group that perform endorphin massage
  Interventions: Other: Endorphin massage
- No interventional Grup 2 (No Intervention): The group that does not perform endorphin massage

INTERVENTIONS:
Other: Endorphin massage — For Group 1 (experimental group), patients admitted to the clinic one day before surgery will complete the first two sections of the Patient Diagnosis Form (I. Individual characteristics and II. Health and illness-related data), the Surgical Fear and Anxiety Scale, and the VAS scales after the endorphin massage. The patients will be informed that the endorphin massage will last approximately 20 minutes. According to evidence-based current guidelines, it is stated that the intensity of the patient's pain should be assessed during the preoperative period for pain management planning and goals in the postoperative period. Therefore, patients' pain scores will also be recorded preoperatively using the VAS scale. On the morning of the surgery, before going to the operating room, the endorphin massage will be repeated, and the scales will be applied again. After surgery, patients will have their pain levels measured using the VAS at hours 0, 4, 8, 16, and 24, and the amount of analgesics tak
  Arms: Endhorphin massage grup

SUMMARY:
This research is planned to investigate the effect of endorphin massage applied before mastectomy surgery on surgical anxiety and fear and pain. This was a randomized, controlled experimental study. The sample comprised 82 patients who underwent mastectomy surgery. This research will be conducted between January 2024 and November 2025 at the Atatürk University Health Practice and Research Hospital, Breast-Endocrine Clinic.The data will be collected using the Introductory Information Form, Surgical Anxiety Scale, Surgical Fear Scale, and Visual Analog Scale.

DETAILED DESCRIPTION:
This research is planned to investigate the effect of endorphin massage applied before mastectomy surgery on surgical anxiety and fear and pain. This was a randomized, controlled experimental study. The sample comprised 82 patients who underwent mastectomy surgery. This research will be conducted between January 2024 and November 2025 at the Atatürk University Health Practice and Research Hospital, Breast-Endocrine Clinic.The data will be collected using the Introductory Information Form, Surgical Anxiety Scale, Surgical Fear Scale, and Visual Analog Scale.

Data Collection The research will be conducted after obtaining institutional permission and ethical committee approval. Following the necessary information provided to the healthcare professionals in the clinic where the study will be conducted, collaboration will be established to carry out the study. Patients who meet the inclusion criteria will be invited to participate after being interviewed one day before the surgery. Verbal and written consent will be obtained from the patients who volunteer and agree to participate in the study. The patients will be divided into two groups according to the randomization list, and all groups will be informed about how to fill out the follow-up forms. In the General Surgery Clinic, mastectomy surgery is scheduled to be performed. Patients are admitted to the clinic one day before the surgery, and if no complications arise, they are discharged on the third day. For pain control, patients will receive pharmacological interventions, including Perfalgan (Paracetamol) 100 ml vial (IV) 2x1, and, if necessary, a weak opioid, Contramal (tramadol hydrochloride) 100 mg (IV). Non-pharmacological interventions for anxiety relief, including pre- and post-surgery education and patient training, will be routinely provided.

Patients in both the experimental and control groups who are admitted to the clinic will be informed about the study, and the researcher will introduce themselves. Patients in the experimental group will be taken to a suitable room for the endorphin massage, where the massage will be applied. During this time, routine preoperative care will be performed by nurses. For Group 1 (experimental group), patients admitted to the clinic one day before surgery will complete the first two sections of the Patient Diagnosis Form (I. Individual characteristics and II. Health and illness-related data), the Surgical Fear and Anxiety Scale, and the VAS scales will be applied after the endorphin massage. The endorphin massage, which will last approximately 20 minutes, will be explained to the patients. The application is in accordance with evidence-based guidelines, which state that the intensity of the patient's pain should be assessed before the surgery for postoperative pain management planning and goals. Therefore, pain scores will be recorded preoperatively using the VAS scale. On the morning of the surgery, before going to the operating room, the endorphin massage will be repeated, and the scales will be applied again. After the surgery, patients will have their pain levels measured using the VAS at hours 0, 4, 8, 16, and 24, and the amount of analgesics taken during the first 24 hours will be recorded.

For Group 2 (control group), no intervention will be applied, and routine preoperative care will be provided by nurses. Before the surgery, without the endorphin massage, the first two sections of the Patient Diagnosis Form, the Surgical Fear and Anxiety Scale, and the VAS scales will be applied to the patients. On the morning of the surgery, the scales will be applied again without any intervention. After surgery, patients will have their pain levels measured using the VAS at hours 0, 4, 8, 16, and 24, and the amount of analgesics taken during the first 24 hours will be recorded.

Key points for Endorphin Massage Application:

The room temperature for the massage should be set between 23-26°C. The massage room should be quiet, with adjustments made to reduce television and monitor sounds, and phones set to silent mode.

The room should be adequately lit. The massage should be given in a position that ensures the patient's comfort.

Randomization:

Due to the nature of the study, the researcher will be involved in the endorphin massage application, data collection, and input stages. Additionally, the women in the intervention group must be informed about the study. Therefore, blinding of the researcher and participants is not possible. However, randomization will be implemented to prevent selection bias. Patients undergoing mastectomy will be screened according to inclusion and exclusion criteria, and eligible participants will be invited to the study. After obtaining written informed consent from those who agree to participate, block randomization will be used to assign participants to two groups. The randomization list will be generated using a computer-based random number table from (https://www.randomizer.org), and participants will be assigned to one of the two groups based on the order of inclusion. Group 1 will consist of patients who receive the endorphin massage, while Group 2 will consist of patients with no intervention.

Data Evaluation Statistical evaluation will be performed using a blinding method. Data analysis will be conducted by a statistician. After ensuring the data is coded and labeled to maintain blinding, the data will be sent to the statistician for analysis. The data will be analyzed using SPSS for Windows 22 software. A statistical significance level of 0.05 will be used, with a Type I error rate of 5% and a 95% confidence interval. Normality distribution of the data will be assessed using Kurtosis and Skewness values (±2). Descriptive statistics such as numbers, percentages, means, and standard deviations will be calculated. For comparisons of the two groups, independent samples t-test will be used for normally distributed measurements, and Mann-Whitney U test will be used for non-normally distributed measurements. For within-group comparisons, dependent samples t-test will be used for normally distributed measurements, and Wilcoxon test will be used for non-normally distributed measurements.

Ethical Principles of the Research

The study will begin after obtaining approval from the Atatürk University Faculty of Medicine Ethics Committee and written permission from the center where the research will be conducted. During data collection, patients will be informed about the study, and the ethical principles of "Informed Consent," "Respect for Autonomy," and "Confidentiality and Protection of Privacy" will be followed. Since individual rights must be protected in the study, the research will adhere to the Helsinki Declaration of Human Rights throughout the study period. Patients who are willing to participate and meet the inclusion criteria will be included in the study. Verbal and written consent will be obtained from the patients before data collection.

Limitations and Generalizability of the Research The study will be limited to patients who are admitted to the Breast-Endocrine Clinic of the Atatürk University Health Practice and Research Hospital, meet the sample selection criteria, and agree to participate. Therefore, the results of the study can only be generalized to patients with characteristics similar to those in this sample group.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above
* Those who are aware of their diagnosis
* Receiving 4-6 cycles of neoadjuvant treatment on a monthly basis
* Scheduled for their first mastectomy surgery
* Those whose cognitive level is suitable for applying the scales

Exclusion Criteria:

* Patients with metastasis
* Patients with a diagnosed severe mental disorder
* Patients enrolled in a different study conducted in the clinic
* Patients who cannot comply with the study process and conditions
* Patients who withdraw from the study at their own request

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 0th hour
  For pain assessment, the patient is asked to indicate the perceived intensity of pain along a 100 mm horizontal line, and this rating is measured starting from the left side. Patients are asked to score their pain level on a scale from 0 to 10 on the horizontal line. 0 represents no pain, and 10 represents unbearable pain. Due to its simplicity, validity, and reliability, this scale is considered the most appropriate tool for describing pain intensity.
Visual Analog Scale (VAS) | 4th hour
  For pain assessment, the patient is asked to indicate the perceived intensity of pain along a 100 mm horizontal line, and this rating is measured starting from the left side. Patients are asked to score their pain level on a scale from 0 to 10 on the horizontal line. 0 represents no pain, and 10 represents unbearable pain. Due to its simplicity, validity, and reliability, this scale is considered the most appropriate tool for describing pain intensity.
Visual Analog Scale (VAS) | 8th hour
  For pain assessment, the patient is asked to indicate the perceived intensity of pain along a 100 mm horizontal line, and this rating is measured starting from the left side. Patients are asked to score their pain level on a scale from 0 to 10 on the horizontal line. 0 represents no pain, and 10 represents unbearable pain. Due to its simplicity, validity, and reliability, this scale is considered the most appropriate tool for describing pain intensity.
Visual Analog Scale (VAS) | 16th hour
  For pain assessment, the patient is asked to indicate the perceived intensity of pain along a 100 mm horizontal line, and this rating is measured starting from the left side. Patients are asked to score their pain level on a scale from 0 to 10 on the horizontal line. 0 represents no pain, and 10 represents unbearable pain. Due to its simplicity, validity, and reliability, this scale is considered the most appropriate tool for describing pain intensity.
Visual Analog Scale (VAS) | 24th hour
  For pain assessment, the patient is asked to indicate the perceived intensity of pain along a 100 mm horizontal line, and this rating is measured starting from the left side. Patients are asked to score their pain level on a scale from 0 to 10 on the horizontal line. 0 represents no pain, and 10 represents unbearable pain. Due to its simplicity, validity, and reliability, this scale is considered the most appropriate tool for describing pain intensity.
Surgical Fear Scale | 1 day before surgery]
  The scale consists of 8 items on a 0-10 numerical scale. This scale, which has two subdimensions, measures the fear related to the short-term and long-term outcomes of the surgical intervention. Items 1-4 assess the fear of the short-term outcomes of the surgery, while items 5-8 measure the fear of the long-term outcomes of the surgery. An increase in the scale score indicates that the fear of surgery is high.
Surgical Fear Scale | On the day of surgery
  : 1 day before surgery]
Surgical Anxiety Scale | 1 day before surgery
  The scale has three subdimensions: Health-Related Anxiety (items 7, 8, 9, 10, 12, and 13), Recovery-Related Anxiety (items 2, 14, 16, and 17), and Procedure-Related Anxiety (items 1, 3, 4, and 5). The total score of the Surgical Anxiety Scale (SAS) is obtained by summing the scores of the subdimension items and the three items not included in any subdimension. The lowest possible score on the scale is 0, and the highest score is 68. As the score increases, the level of surgical anxiety is considered higher.
Surgical Anxiety Scale | On the day of surgery]
  The scale has three subdimensions: Health-Related Anxiety (items 7, 8, 9, 10, 12, and 13), Recovery-Related Anxiety (items 2, 14, 16, and 17), and Procedure-Related Anxiety (items 1, 3, 4, and 5). The total score of the Surgical Anxiety Scale (SAS) is obtained by summing the scores of the subdimension items and the three items not included in any subdimension. The lowest possible score on the scale is 0, and the highest score is 68. As the score increases, the level of surgical anxiety is considered higher.

CONTACTS AND LOCATIONS:
Overall Officials: MERVE KAYA, Principal Investigator — Ataturk University

IPD SHARING:
Plan to Share IPD: No